CLINICAL TRIAL: NCT02174458
Title: Outcome in Body Contouring Surgery After Major Weight Loss - a Prospective Matched Single Blind Study
Brief Title: Body Contouring Surgery After Massive Weight Loss
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: BC_QoL_EK_311/13
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Weight Loss
Keywords: Bariatric surgery; Body contouring; Quality of life
MeSH Terms: conditions — Weight Loss | interventions — Body Contouring

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bariatric Surgery only: Patients after Bariatric Surgery but no secondary reconstructive procedures
- Body Contouring surgery: Post-bariatric patients and patients with no history of bariatric surgery but after natural weight loss
  Interventions: Procedure: Body Contouring Surgery

INTERVENTIONS:
Procedure: Body Contouring Surgery — Patients after bariatric surgery (BS) and patients with no history of BS but after natural weight loss and some degree of skin laxity who underwent Body contouring will be included after written informed consent is obtained.
  Other Names: Body Contouring Surgery is the excision of excess skin
  Groups: Body Contouring surgery

SUMMARY:
Body contouring (BC) surgery after major weight loss (MWL) requires extensive and multiple procedures. Yet, there are inconsistent data regarding the outcome after BC procedures. The aim of this study is to investigate the outcome from patients who elect to have BC procedures after MWL treated at a single metropolitan tertiary referral center.

DETAILED DESCRIPTION:
Background The obesity epidemic worldwide continues to worsen, with rates in Europe and North America estimated at about 20-30% of the adult population.(Vico et al., 2010) It is defined as a body mass index (BMI) above 30, and morbid obesity as a BMI above 40kgm-2.(Strauch et al., 2006; Vico et al., 2010) As a consequence, there is an explosive growth of obesity-associated comorbidities, associated with high healthcare costs.(Reiffel et al., 2013) One of the few consistent means of achieving a significant weight-loss in morbidly obese patients is bariatric surgery (BS).(Buchwald et al., 2004; Maggard et al., 2005) Shermak et al. defined massive weight loss (MWL) as 50% or greater loss of excess weight.(Shermak et al., 2006) Next to the amelioration of the medical comorbidities associated with obesity, patients also benefit from improvement in their psychosocial functioning, personal health perceptions and health-related quality of life.(Karlsson et al., 1998; Karlsson et al., 2007; Sarwer et al., 2008) A major drawback after BS is the persistence of large quantities of excess and inelastic skin and subcutaneous tissue. Thus, patients often experience skin irritations, mycotic infections and secondary self-imaging problems.(Reiffel et al., 2013; Vico et al., 2010) Body contouring (BC) surgery, usually excisional, includes (circumferential) abdominoplasty, breast reduction, panniculectomy, brachioplasty, and thigh lift. It removes the excess tissue which remains after massive weight loss and consecutively leads to a significant improvement in self-image and self-esteem, as well as mobility, overall daily functioning and hygiene.(Larsen et al., 2007; Song et al., 2006) These procedures are usually multiple and extensive. Thus, combining and reducing the number of such procedures while obtaining optimal results would be most beneficial to both the surgeon and the patient.(Ellabban and Hart, 2004; Hallock and Altobelli, 1985) For patients who seek BS, quality of life is an important issue. In a recent study by Modarressi et al. it has been shown that Roux-en-Y gastric bypass (RYGBP) improves the health-related quality of life (HRQoL). Furthermore, it was shown that HRQoL is directly related to weight loss and BC procedures further improves HRQoL in comparison to RYGBP alone, as evidenced by the Moorehead-Ardelt questionnaire.(Modarressi et al., 2013; Oria and Moorehead, 1998) Nevertheless, there is an urgent need to develop specific and well-constructed patient reported outcome (PRO) instruments in order to obtain reliable information regarding QoL and patient satisfaction following BC surgery in MWL patients.(Jabir, 2013)

Clinical Data In the literature there are some inconsistent data regarding QoL scales after BC procedures.(Singh et al., 2012) Problems after MWL with excessive skin folds compromises body image and may negatively impact the physical and mental components of QoL.(Mitchell et al., 2008) Thus, theoretically, after removal of skin excess, the QoL scales should improve after BC procedures. Indeed, several studies have demonstrated improvements in QoL associated with BC surgery.(Coriddi et al., 2011; Pecori et al., 2007; Song et al., 2006; van der Beek et al., 2010) However, in a recent study by Singh et al., scales comprising the mental component were lower in the group of patients who received BC procedures, indicating impaired QoL.(Singh et al., 2012) Of those, role-emotional and social functioning were significantly lower than both the control and the post-bariatric surgery group, showing that those patients who elected to have BC procedures suffer from worsening inhibited social interactions.(Singh et al., 2012) It might be arguable that patients in the post-bariatric surgery group who elected not to undergo BC chose so because their QoL was already high.(Singh et al., 2012) Thus, counseling and education prior to plastic surgery is extremely important to ensure appropriate expectations for the patient in regard to scarring and the realistic scope that can be accomplished by surgery.(Singh et al., 2012) QoL, especially in women aged between 35 to 64 years old, is the most affected domain in patients with BMI > 40kg/m2.(Larsson et al., 2002) This dissatisfaction motivates different behaviours, including exercise, weight loss and cosmetic surgery.(Sarwer et al., 2008) Thus, despite obesity is more prevalent in men, it might explain partially why women more frequently seek bariatric surgery.(Modarressi et al., 2013) Following BS, patients are initially enthusiastic to see cure of their diabetes, decreased pain in their joints and weight loss.(Colwell, 2010) Nevertheless, the skin does not contract with the volume loss.(Colwell, 2010) As soon as the weight has been stable for at least 6 months, plastic surgical evaluation seems to be appropriate.(Colwell, 2010) In general, the lower the BMI at the time of BC surgery, the better the result.(Langer et al., 2011) Usually, condouting procedures are preserved for those patients who attain a BMI less than or equal to 35.(Arthurs et al., 2007) To date, little is known about the frequency and proportions of patients who undergo BS and consequently receive BC surgery. Reasons for not undergoing body contouring procedures can be the lack of awareness regarding options and expense.(Reiffel et al., 2013) Documentation of functional problems, such as rashes, sexual dysfunction and difficulty with exercise are important in attempting to obtain insurance coverage for at least part of their surgery.(Arthurs et al., 2007) Panniculectomy, defined as removal of excess skin and fat in the abdomen without umbilical transpostion, is the surgical procedure most likely to be covered by insurance.

Usually, truncal deformity is the most common presenting complaint of MWL patients, and the procedure of choice is a lower body lift.(Colwell, 2010) It is crucial to focus postoperatively on patient safety prioritizing in seroma prevention and deep vein thrombosis (DVT) prophylaxis. Reported complication rates postoperative range between 17-50% including wound-healing problems, haematoma, infection, necrosis or pulmonary embolism.(Vico et al., 2010) Furthermore, many of these patients have psychiatric problems, and thus counseling, especially in the perioperative period is extremely important.(Langer et al., 2011) The number of procedures that can safely be performed in one sitting depends on the patient's anatomy, the surgeon, the surgical facility and overall medical health.(Arthurs et al., 2007) The patient's BMI should be normal or slightly overweight. Otherwise, staging the procedures into two or more surgeries separated by 3-6 months is suggested.(Arthurs et al., 2007) Ideally, the operative time should be kept under six hours or below to minimize complications.(Langer et al., 2011) Obviously, if vectors of pull at surgery are in opposite directions, such as in an upper body lift and a belt lipectomy/lower body lift, these procedures should be performed separately.(Langer et al., 2011) In a study by Ellabban et al., 14 patients were evaluated who underwent BC operations using combined abdominoplasty and medial thigh reduction. The authors concluded that combined abdominoplasty with vertical medial thigh reduction is effective in correcting aesthetic and physical problems after massive weight reduction with an excellent predictable outcome.(Ellabban and Hart, 2004) Also, combined brachioplasty, thoracoplasty, and mammoplasty has proven to be safe, effective, and beneficial for both the surgeon and patient.(Hallock and Altobelli, 1985) In order to establish an evidence base to support the idea that BC is as much (or even more) a functional procedure as it is cosmetic, a flurry of studies assessing QoL and patient satisfaction following BC surgery has been resulted.(Jabir, 2013) The method of choice to assess QoL and patient satisfaction is to use patient specific psychometrically validated PRO measures.(Jabir, 2013) To date, none of the measures have been specifically developed for BC surgery patients. Instead, there is an urgent need to develop specific and well- constructed PRO instruments in order to obtain reliable information regarding QoL and patient satisfaction after BC surgery in MWL patients.(Jabir, 2013)

STUDY OBJECTIVES The main objective of this research is to analyse QoL and patient satisfaction after BC surgery in MWL male and female patients.

We hypothesize that >80% of the patients have a total score of +2.25 to +3 ("much better") or +0.75 to +2 ("better") in the Moorehead-Ardelt questionnaire. 66 patients of equal distribution and demographic characteristics after bariatric surgery but no secondary reconstructive procedure will serve as a control group.

The associated research questions are as follows:

What is the outcome in patients after BC surgery and MWL concerning:

Hypotheses:

Primary outcome:

After a mean follow-up of 8.9±3.5 years after BC surgery we hypothesize that >90% of the 66 patients will answer the survey. Based on the literature(Modarressi et al., 2013), we expect that >80% of the patients have a total score of +2.25 to +3 ("much better") or +0.75 to +2 ("better") in the Moorehead-Ardelt questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Weight loss > 15kg
* Age > 18 years

Exclusion Criteria:

* Weight loss < 15kg
* Age < 18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-bariatric male and female patients and patients with no history of bariatric surgery but after natural weight loss and some degree of skin laxity who underwent body-contouring surgery between February 1999 and October 2009 at the Department of Plastic, Reconstructive and Aesthetic Surgery, Handsurgery, University Hospital of Basel will be included. Patients after BS with equal distributions and demographic characteristics but no secondary reconstructive procedures served as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Quality of life after Body contouring Surgery | 10 years
  The Moorehead-Ardelt(Oria and Moorehead, 1998) questionnaire is the HRQoL part of the "Bariatric Analysis and Reporting Outcome System". This questionnaire was created to specifically evaluate the outcome of bariatric surgery, and it is widely used by national and international bariatric surgery associations. It evaluates five domains of HRQoL: self-esteem, physical activity, social life, work ability and sexual activity. For each domain, patient evaluates "much better", "better", "same", "worse" or "much worse" his status on the time that he answers to the questionnaire in comparison to his status before bariatric surgery. Results are summarized in a total score (-3.0 to +3.0) which is the sum of the self-esteem score (-1 to +1) and the four other domains (-0.5 to +0.5 for each). Total score is estimated as "much better" (scores +2.25 to +3), "better" (+0.75 to +2), "same" (+0.5 to -0.5), "worse" (-0.75 to -2 points) and "much worse" (-2.25 to -3).(Modarressi et al., 2013)

SECONDARY OUTCOMES:
Comparison of the sub-Domains of the Moorehead-Ardelt questionnaire after Body Contouring Surgery | 10 Years
  Comparisons between the five domains of the Moorehead-Ardelt questionnaire Drop-out rate

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Kalbermatten, MD, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Basel, Switzerland